CLINICAL TRIAL: NCT03917563
Title: Registry to Evaluate Chinese Real-World Clinical Outcomes in Patients With AF Using the WATCHMAN Left Atrial Appendage Closure Technology
Acronym: RECORD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Hospital (Other Government); the PLA General Hospital (Unknown); Beijing Chao Yang Hospital (Other); Peking University First Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai 10th People's Hospital (Other); Changhai Hospital (Other); Dongfang Hospital Affiliated to Tongji University (Other); Shanghai 6th People's Hospital (Other); Ruijin Hospital (Other); Shanghai Thoracic Hospital (Unknown); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shenzhen Sun Yat-sen Cardiovascular Hospital (Other); Tianjin Medical University General Hospital (Other); Southwest Hospital, China (Other); Shengjing Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Central Hospital of Dalian (Unknown); General Hospital of Shenyang Military Region (Other); Qilu Hospital of Shandong University (Other); The Second Hospital of Hebei Medical University (Other); Shanxi Cardiovascular Hospital (Other); People's Hospital of Taizhou (Unknown); The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Ningbo No. 1 Hospital (Other); Sir Run Shaw Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan Asia Heart Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); General Hospital of Ningxia Medical University (Other); Sichuan Provincial People's Hospital (Other); West China Hospital (Other); ZhuHai Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20182078-X-1
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): WATCHMAN LAA occluder treatment
  Interventions: Device: WATCHMAN LAA occluder

INTERVENTIONS:
Device: WATCHMAN LAA occluder — WATCHMAN LAA occluder

SUMMARY:
The aim of the registry is to evaluate Chinese real-World clinical outcomes in patients With AF using the WATCHMAN left Atrial appendage closure technology

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or above;
2. Patient is eligible for a WATCHMAN device according to current international and local guide-lines and per physician discretion;
3. Patient is willing and capable of providing informed consent to participate in all procedures associated with receiving a WATCHMAN device at an approved clinical investigational center.

Exclusion Criteria:

1. Patient is currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments.
2. Patient is a woman of childbearing potential who is, or plans on becoming, pregnant during the duration of follow-up assessments required as part of the WATCHMAN procedure.
3. Patient is unable or not willing to complete follow-up visits and examination as required as part of the WATCHMAN procedure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2019-04-20 (Estimated); Primary Completion 2021-04-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
The composite primary endpoint of the stroke, systemic embolism, or cardiovascular or unexplained death | 12 months post procedure

SECONDARY OUTCOMES:
Bleeding | Periprocedure and 1,5,6, 12, 24, 36, 48, 60 month post procedure
  Life threatening or disabling, major bleeding and Minor bleeding
Vascular access-related complications | Periprocedure and 1,5,6, 12, 24, 36, 48, 60 month post procedure
  Haematoma at access site<6 cm; Retroperitoneal haematoma;Arteriovenous fistula;Vascular surgical repair at catheter access sites;Pulmonary embolism;Ipsilateral deep vein thrombosis;Access site-related infection requiring intravenous antibiotics or extended hospitalization
Device-related complications | Periprocedure and 1,5,6, 12, 24, 36, 48, 60 month post procedure
  Device embolization; Device erosion;Clinically significant device interference with surrounding structure;Device thrombus;Device fracture;Device infection/endocarditis/pericarditis;Device perforation/laceration;Device allergy

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, Principal Investigator — Xijing Hospital
Locations (1):
- Ling Tao, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gao C, Su F, Liu J, Zhang T, Ning Z, Yang B, Chu H, He B, Zhang J, Zhou L, Li Y, Zhang Y, Hu H, Xu Y, Zeng J, Guo J, Su X, Ruan ZB, Liu H, Wang P, Garg S, Soliman O, Holmes DR Jr, Serruys PW, Tao L; RECORD Investigators. 1-Year Clinical Outcomes and the Impact of Procedural Configurations in Left Atrial Appendage Occlusion Patients. JACC Asia. 2024 Oct 1;4(10):777-790. doi: 10.1016/j.jacasi.2024.07.013. eCollection 2024 Oct. PMID 39553900